CLINICAL TRIAL: NCT00425230
Title: Pilot Study of Use of Duloxetine for the Treatment of Phantom Limb Pain
Brief Title: Open Label Study of Duloxetine for the Treatment of Phantom Limb Pain
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: No patients were enrolled in this study. The study onset was delayed due to problems with drug acquisition.
Sponsor: Baylor College of Medicine (Other)
Responsible Party: Principal Investigator, Wayne Goodman MD, Chair/Professor, Baylor College of Medicine
Allocation: Non-Randomized | Model: Single Group | Masking: None
Other Study IDs: H-19539
Record Dates: First submitted 2007-01-19; First posted 2007-01-22 (Estimated); Last update posted 2022-08-12 (Actual); Status verified 2022-08

CONDITIONS: Chronic Phantom Limb Pain
MeSH Terms: interventions — Duloxetine Hydrochloride

INTERVENTIONS:
Drug: Duloxetine

SUMMARY:
This is a study to assess the possible benefit of duloxetine in the treatment of chronic phantom limb pain.

ELIGIBILITY:
Inclusion Criteria:

1. Chronic PLP > 6 months
2. Short-Form McGill Pain Questionnaire Sensory Pain Rating Index raw score ≥ 16
3. Age ≥ 18 years old
4. Inpatient or Outpatient
5. Able to come to all appointments, in the opinion of the investigator
6. Able to give informed consent, in opinion of investigator

Exclusion Criteria:

1. Current Major Depressive disorder, Anxiety Disorder, or Psychotic disorder assessed by the Mini International Neuropsychiatric Interview (MINI)
2. Substance abuse or dependence within the last six months, as assessed by the MINI
3. Known Diabetes Mellitus to exclude diabetic peripheral neuropathy
4. History of coronary artery disease, hepatic disease, renal disease
5. Other pain syndromes
6. Any unstable medical conditions in the opinion of the investigator
7. Other psychotropic medications excluding hypnotics

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 15 (Estimated)
Dates: Start 2007-01; Study Completion 2007-06

PRIMARY OUTCOMES:
McGill Short Form Pain Questionairre

SECONDARY OUTCOMES:
Fiser Side effect scale
visual analog pain scale
Present Pain intensity
Tylenol # 3 consumption

CONTACTS AND LOCATIONS:
Overall Officials: Asif Chaudhry, MD, Principal Investigator — Baylor College of Medicine
Locations (1):
- Micheal E. DeBakey Veterans Hospital, Houston, Texas, United States